CLINICAL TRIAL: NCT00062894
Title: A Multi-Center Study to Examine the Pharmacokinetics, Whole Body and Organ Dosimetry, and Biodistribution of Fission-Derived Iodine I 131 Tositumomab for Patients With Previously Untreated or Relapsed Follicular or Transformed Follicular Non-Hodgkin's Lymphoma
Brief Title: Study of Untreated or Transformed Follicular Non-Hodgkin's Lymphoma With Fission-Derived Iodine I 131 Tositumomab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCBX001-048
Record Dates: First submitted 2003-06-17; First posted 2003-06-19 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-09

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Iodine I 131 Tositumomab; BEXXAR; non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

INTERVENTIONS:
Drug: Iodine I 131 Tositumomab

SUMMARY:
The purpose of this study is to assess the blood pharmacokinetics in patients with previously untreated or relapsed follicular or transformed follicular non-Hodgkin's lymphoma who have received a dosimetric dose of fission-derived iodine I 131 tositumomab.

DETAILED DESCRIPTION:
This is a multi-center study in which 12 patients with previously untreated or relapsed follicular or transformed follicular non-Hodgkin's lymphoma will receive a dosimetric dose of fission-derived Iodine I 131 Tositumomab followed by a therapeutic dose of tellurium-derived Iodine I 131 Tositumomab. Blood Pharmacokinetics, total body clearance, tumor and organ dosimetry, and biodistribution will be assessed following administration of the dosimetric dose.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Histologically confirmed diagnosis of follicular lymphoma, Grade 1, 2, or 3, or diffuse large cell lymphoma (WHO/REAL classification).

Follicular, small cleaved; Follicular, mixed small cleaved and large cell; Follicular large cell lymphoma Transformed diffuse large cell lymphoma following or concurrent with a diagnosis of follicular lymphoma.

* Stage III or IV disease at the time of study entry.
* Previously untreated or recurrent lymphoma after no more than four prior qualifying therapy regimens.
* Performance status of at least 70% on the Karnofsky Performance Scale and an anticipated survival of at least three months.
* Bi-dimensionally measurable disease with at least one lesion measuring greater than or equal to 2.0 cm x 2.0 cm (=4.0 cm2)by CT scan.
* Absolute B lymphocyte count (as determined by CD 19 reactivity)of 30 to 350 cell/mm3 within 21 days prior to study enrollment.
* ANC greater than or equal to 1500 cells/mm3; absolute lymphocyte count within normal limits; and platelet count greater than or equal to 150,000/mm3 within 21 days prior to study enrollment. Blood products and/or growth factors should not have been taken within 4 weeks prior to blood draw.
* Adequate renal function (defined as serum creatinine < 1.5 x ULN) and hepatic function (defined as total bilirubin < 1.5 x ULN and AST < 5 x ULN) within 21 days of study enrollment.
* Human Anti-Murine Antibody (HAMA) negative within 21 days prior to study enrollment.
* Signed IRB approved consent form prior to any study-specific procedures being implemented.

Exclusion Criteria:

* Greater than 25% of the intratrabecular marrow space involved by lymphoma in bone marrow biopsy specimens as assessed microscopically within 90 days of study enrollment. Bilateral posterior iliac crest core biopsies are required if the core obtained on a unilateral biopsy is less than 2 cm.
* Prior chemotherapy, biologic therapy, steroids, or radiation therapy as treatment for their NHL within 28 days prior to study enrollment.
* Prior Rituximab therapy within 120 days prior to study enrollment.
* Prior radioimmunotherapy.
* Prior splenectomy.
* Splenomegaly defined as spleen mass greater than 700 grams.
* Bulky disease as defined as any unidimensional measurement of lymphomatous mass exceeding 7 cm.
* Prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the patient has a generally accepted risk of recurrence less than 20%.
* Central nervous system involvement by lymphoma.
* Evidence of active infection requiring IV antibiotics at the time of study enrollment.
* Known HIV infection.
* New York Heart Association class III or IV heart disease or other serious illness that would preclude evaluation.
* Active obstructive hydronephrosis.
* Evidence of clinically significant ascites or pleural effusion observed on screening physical exam or baseline CAT xcan.
* Prior myeloablative therapy.
* History of failed stem cell collection.
* Pregnant or nursing patients. Patients of childbearing potential must undergo a serum pregnancy test within 7 days of study enrollment and radiolabeled antibody is not to be administered until a negative result is obtained. Males and females of childbearing age, must agree to use effective contraception for six months following the radioimmunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-04; Study Completion 2007-04

PRIMARY OUTCOMES:
To assess the blood pharmacokinetics in patients with previously untreated or relapsed follicular or transformed follicular non-Hodgkin's lymphoma

SECONDARY OUTCOMES:
12 patients with previously untreated or relapsed follicular or transformed follicular non-Hodgkin's lymphoma will receive a dosimetric dose of fission-derived Iodine I 131 Tositumomab

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - Bay Pines VA Medical Center, Bay Pines, Florida
  - Rush Medical Center, Chicago, Illinois
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania